CLINICAL TRIAL: NCT00546728
Title: The Chronic and Acute Postprandial Vascular Effects of Exenatide vs. Metformin in Abdominally Obese Patients With Impaired Glucose Tolerance
Brief Title: The Vascular Effects of Exenatide Versus Metformin in Patients With Pre-Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Paul Heart Clinic (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry); Eli Lilly and Company (Industry); International Diabetes Center at Park Nicollet (Other)
Responsible Party: Principal Investigator, Aaron S. Kelly, Ph.D., Assistant Professor, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHC 2007-02
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-09

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Exenatide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): Subjects were randomlly assigned to treatment arm: Exenatide 10 mcg twice daily vs. Metformin 500 mg twice daily.
  Interventions: Drug: Exenatide
- Metformin (Active Comparator): Subjects were randomlly assigned to treatment arm: Exenatide 10 mcg twice daily vs. Metformin 500 mg twice daily.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Exenatide — exenatide 10 mcg twice daily
  Arms: Exenatide
Drug: Metformin — metformin 500 twice daily
  Arms: Metformin

SUMMARY:
The purpose of this study is to compare the effects of exenatide versus metformin on vascular health with chronic (3-month) therapy and during a 2-hour period following a meal in patients with pre-diabetes. It is predicted that exenatide will improve vascular health to a greater degree compared to metformin.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years old
* Impaired glucose tolerance: 2-hr oral glucose tolerance test (OGTT) plasma glucose >140 mg/dL OR impaired fasting glucose: fasting glucose > or = 100 mg/dL OR elevated glycosylated hemoglobin: Hemoglobin A1c > or = 5.7%
* Abdominal obesity: waist circumference >102 cm (men) and >88 cm (women)
* Stable cardiovascular medication regimen (or other medications known to affect endothelial function) at least 1 month prior to enrollment and throughout the study

Exclusion Criteria:

* Type 2 diabetes
* Current use of glycemic control medications within one month of randomization
* Fasting glucose >126 mg/dL
* Current use of weight loss medication
* Previous weight loss surgery
* History of severe gastrointestinal disease
* Standard clinical contraindications to exenatide or metformin therapy
* Unstable angina
* Heart failure
* Stroke or coronary artery bypass graft within 3 months of screening
* Women who are currently pregnant or planning to become pregnant
* Breastfeeding women
* Clinically significant liver disease
* Creatinine > 1.5 mg/dL
* Hepatic function greater than 3 times upper limit of normal
* Patients who are mentally incompetent and cannot sign a Patient Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S. Kelly, Ph.D., Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - International Diabetes Center at Park Nicollet, Saint Louis Park, Minnesota
  - St. Paul Heart Clinic, Saint Paul, Minnesota

REFERENCES:
- [Derived] Kelly AS, Bergenstal RM, Gonzalez-Campoy JM, Katz H, Bank AJ. Effects of exenatide vs. metformin on endothelial function in obese patients with pre-diabetes: a randomized trial. Cardiovasc Diabetol. 2012 Jun 8;11:64. doi: 10.1186/1475-2840-11-64. PMID 22681705

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from medical clinics
Groups:
- Exenatide: Three months of Exenatide. Exenatide was initiated at a dose of 5 mcg, twice a day for one month and up titrated to 10 mcg, twice a day for the remaining two months.
- Metformin: Three months of Metformin. Metformin was initiated at a dose of 500 mg, twice a day for one month and up titrated to 1000 mg, twice a day for the remaining two months.
Period: Overall Study
Arm/Group | Exenatide | Metformin
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exenatide: Three months of Exenatide therapy. Exenatide was initiated at 5 mcg, twice a day for one month and then up titrated to 10 mcg, twice a day for the remaining two months.
- Metformin: Three months of Metformin therapy. Metformin was initiated at 500 mcg, twice a day for one month and then up titrated to 1000 mcg, twice a day for the remaining two months.
- Total: Total of all reporting groups
Arm/Group | Exenatide | Metformin | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10) | 58.4 (10.1) | 58.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Reactive Hyperemic Index Over the 3-month Treatment Period
Description: Change in reactive hyperemic index over the 3-month treatment period, which is a measure of endothelial (inner lining of blood vessels) function. This is measured as a ratio of post-occlusion blood flow volume versus baseline blood flow volume in fingertips. Higher ratio values are considered indicative of better arterial health.
Time Frame: Change from baseline to 3 months
Population: All completers were included in the analysis
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Exenatide | Metformin
Number analyzed (Participants) | 25 | 25
ratio | 0.01 (0.68) | -0.17 (0.72)

ADVERSE EVENTS:
Time Frame: 3-months
Arm/Group | Exenatide | Metformin
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
unblinded study design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No